CLINICAL TRIAL: NCT00652067
Title: IND for One Patient to Receive Clofazamine for Treatment of MAI
Brief Title: Clofazamine for the Treatment of Mycobacterium Avium Intracellulare(MAI)
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Margaret Pisani, MD, Yale University School of Medicine
Other Study IDs: 0604001371
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Infection, Mycobacterium Avium-Intracellulare
Keywords: Mycobacterium avium-intracellulare
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Only one patient is being treated under a single patient IND.

SUMMARY:
This protocol is an single patient IND to provide clofazamine to treat one patient who has MAI and is resistant to or can not tolerate standard of care. The drug is not otherwise available.

ELIGIBILITY:
Inclusion Criteria:

* Treatment of one patient with MAI

Exclusion Criteria:

* No other patients will be treated

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Single patient
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Pisani, M.D., Principal Investigator — Yale University